CLINICAL TRIAL: NCT00392483
Title: The Use and Diffusion of an E-learning Programme in Diagnostic Evaluation of Dementia Among General Practitioners in Denmark
Brief Title: Reuptake of an E-Learning Programme in General Practice
Status: Completed | Type: Observational
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Other Study IDs: CHP-06-02-FEAP
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2006-11

CONDITIONS: Education; Dementia
Keywords: Heading Health Plan Implementation; Computer-Assisted Instruction; General Practice; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The evaluate the use and diffusion of an E-learning programme in Diagnostic Evaluation of Dementia among General Practitioners (GPs) in Denmark.

The hypothesis are:

1. The GPs do not use the guided instructions
2. The GPs using the programme are more frequently younger GPs.
3. GPs working in rural areas will use the programme more frequently

DETAILED DESCRIPTION:
In a period from november 2006 to may 2007 all log files of those GPs who log on to the E-learning programme are kept by the Danish Medical Association. They are handed over to the principal investigator in an anonymous form.

ELIGIBILITY:
GPs stopping working as GPs in study period

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All GPs in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 3632 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans B Waldorff, PhD, Principal Investigator — Research Unit of General Practice
Locations (1):
- Research Unit of General Practice, Copenhagen, Capital, Denmark

REFERENCES:
- [Result] Waldorff FB, Steenstrup AP, Nielsen B, Rubak J, Bro F. Diffusion of an e-learning programme among Danish General Practitioners: a nation-wide prospective survey. BMC Fam Pract. 2008 Apr 25;9:24. doi: 10.1186/1471-2296-9-24. PMID 18439279